CLINICAL TRIAL: NCT06918041
Title: FiberLocker® System Augmentation of Rotator Cuff Repairs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ZuriMED Technologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZM102024
Record Dates: First submitted 2025-03-06; First posted 2025-04-09 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Rotator Cuff Tear; Rotator Cuff Tears; Rotator Cuff Tears of the Shoulder
Keywords: Rotator Cuff Tears; Rotator Cuff Repair; Augmentation; Reinforcement; Mechanical Augmentation; Rotator Cuff Degeneration
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Augmentation of Rotator Cuff Repair using the FiberLocker® System (Experimental): All enrolled participants will undergo repair of the rotator cuff tear, with augmentation utilizing the FiberLocker® System.
  Interventions: Device: FiberLocker® System (encompassing FiberLocker® Instrument SN & SpeedPatch® PET)

INTERVENTIONS:
Device: FiberLocker® System (encompassing FiberLocker® Instrument SN & SpeedPatch® PET) — The FiberLocker® System is a mechanical augmentation system that includes an implant (SpeedPatch® PET) and an instrument (FiberLocker® Instrument SN) for its attachment. The implant is composed of non-woven PET fibers, and the instrument features a reciprocating needle at its tip, which pushes the individual patch fibers into the underlying tendon tissue.

SUMMARY:
The purpose of this study is to prospectively evaluate healing, functional clinical outcomes, and safety of arthroscopic rotator cuff repairs augmented with the FiberLocker® System (encompassing the SpeedPatch® PET and the FiberLocker® Instrument SN).

The primary outcome measure is healing evaluation based on Magnetic Resonance Imaging (MRI) at a minimum of 6 months post-operatively.

The secondary outcome measures are the Sugaya classification, Goutallier Stage and tendon quality based on MRI as well as objective scores and patient-reported outcome measures (PROMs) from validated outcome scoring systems.

ELIGIBILITY:
Inclusion Criteria:

1. The Subject is between the ages of 30 and 70 years.
2. Subject is planning to undergo arthroscopic surgery for full-thickness rotator cuff tear (RCT)
3. Tear size ≥ 2 cm
4. Primary rotator cuff repair
5. Subject preoperative MRI obtained within 1 year prior to surgery

Exclusion Criteria:

1. The Subject is unable or unwilling to sign the Patient Informed Consent, approved by the Institutional Review Board.
2. The Subject objects to the use of the FiberLocker® System
3. History or known allergy or intolerance to polyester
4. Complete full-thickness subscapularis tears of > than the superior 1/3 of the tendon (Lafosse grade 3 and above)
5. Hamada grade III and above
6. Less than 2 mm joint space of the glenohumeral joint on either an anteroposterior or axillary radiograph
7. Recurrent shoulder instability
8. Corticosteroid injection in the operative shoulder within three months before surgery
9. Subjects with inflammatory or auto-immune based joint diseases (e.g., rheumatoid arthritis, systemic lupus erythematosus)
10. Subjects with current acute infection in the area surrounding the surgical site
11. Revision rotator cuff repair
12. Pregnant or planning to become pregnant during the study period
13. Subject is breastfeeding during the study period
14. Subject has conditions or circumstances that would interfere with study requirements

Intraoperative Exclusion Criteria:

1. Partial rotator cuff repairs
2. Lafosse grade 3 or higher subscapularis tears
3. Limited space for implant delivery
4. FiberLocker® System cannot be used as indicated

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Healing Evaluation | Pre-operatively & minimum 6 months post-operatively
  The primary outcome measure is healing evaluation based on Magnetic Resonance Imaging (MRI) at a minimum of 6 months post-operatively.
  A standard shoulder MRI protocol utilizing a minimum of a 1.5 Tesla magnet will be utilized. The cuff integrity will be classified using the 5 categories described by Sugaya et al. Thereby, type IV and V are considered as retear and type I, II, and III as healed. The healing rate will be estimated and reported descriptively, and a 95% confidence interval will be reported assuming a binomial distribution (unless otherwise noted).

SECONDARY OUTCOMES:
Sugaya Classification | Minimum 6 months post-operatively
  The Sugaya Classification based on MRI images is used to evaluate the integrity of a repaired rotator cuff and to assess healing outcomes after a repair. The classification uses a categorial scoring system with grades from Type I to Type V. - Type I: Normal thickness and low signal intensity in all sections
  * Type II: Normal thickness and high signal intensity
  * Type III: Insufficient thickness without discontinuity, representing a partial-thickness tear
  * Type IV: Minor discontinuity (1-2 slices) on both oblique coronal and oblique sagittal images
  * Type V: Major discontinuity (>2 slices) on both oblique coronal and sagittal images
Goutallier Stage | Pre-operatively & minimum 6 months post-operatively
  The Goutallier Classification is evaluated using MRI images to assess fatty infiltration and muscle degeneration in the rotator cuff. It has a categorial grading system from stage 0 to 4.
  Based on MRI images, the investigator classifies the rotator cuff of each subject. Thereby, a higher classification means more fatty infiltration.
Tendon Quality | Pre-operatively & minimum 6 months post-operatively
  The tendon quality of each subject is graded based on MRI images using a categorial scoring system.
  The following classification can be used: Normal, Intact with edema/regularity, Partial tearing and/or abnormal tissue, Complete Tear/Abnormal.
American Shoulder and Elbow Surgeons (ASES) Score | Pre-operatively, Post-operatively: 6 months, 12 months, 24 months
  The ASES score is a patient-reported outcome measure survey which is completed by all subjects. It is used to assess shoulder function and pain. Based on the answers, a final score between 0 and 100 can be achieved. Thereby, higher scores indicate better shoulder function and less pain.
Single Assessment Numeric Evaluation (SANE) Score | Pre-operatively, Post-operatively: 6 months, 12 months, 24 months
  The SANE score is a patient-reported outcome measure used to assess a patient's perception of their shoulder function. It consists of a single question and each subject has to rate their shoulder function on a scale from 0% to 100%. Thereby, higher percentages indicates better shoulder function.
Visual Analog Scale for pain (VAS Score) | Pre-operatively, Post-operatively: 2 weeks, 6 months, 12 months, 24 months
  The VAS Score is a patient-reported outcome measure used to assess pain intensity. All patients rate their pain on a horizontal line ranging from 0 to 10. Thereby, a higher score indicates greater pain intensity.
Veterans RAND 12-Item Health Survey (VR-12) | Pre-operatively, Post-operatively: 6 months, 12 months, 24 months
  The VR-12 is a patient-reported outcome measure assessing physical and mental health of the subjects. Based on their answers, the subjects can reach a score between 0 and 100, with a higher score indicating better health.
Range of Motion (ROM) Assessment | Pre-operatively, Post-operatively: 6 months, 12 months, 24 months
  The subject's active ROM (based on the objective ASES score) is assessed using a goniometer. During an outpatient visit at the investigators facility, forward flexion, external rotation, abducted external rotation, abducted internal rotation and internal rotation will be evaluated. The unit of measure is degrees.
  If subjects are unable to return for an in person visit, an optional self-assessment of these range of motion form will be provided for electronic completion.
Strength Assessment | Pre-operatively, Post-operatively: 6 months, 12 months, 24 months
  The strength of each subject will be evaluated (based on objective ASES) using a manual muscle testing device or other dynamometers. Thereby, external rotation strength, subscapularis strength-belly press and the constant score strength will be evaulated. The unit of measure will be kilograms or pounds.
Constant-Murley Score | Pre-operatively, Post-operatively: 6 months, 12 months, 24 months (all optional)
  The Constant-Murley Score will be assessed optionally. The score requires an outpatient visit at the investigator's facility and covers questions and functional assessments to assess pain, activity levels, range of motion and strength. The range of motion is assessed using a goniometer in degrees and the strength using a manual muscle testing device (or other dynamometers) in kilogram. The subjects can reach points between 0 and 100, whereby a higher score indicates better function.
(Serious) Adverse Events, (Serious) Adverse Device Effects and Device Deficiencies | From the surgical intervention to 24 months postoperatively
  (Serious) Adverse Events, (Serious) Adverse Device Effects and Device Deficiencies will be reported by the research staff as soon as they occur.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Rush University Medical Center, Chicago, Illinois
  - MedStar Health Research Institute, Columbia, Maryland
  - Wake Forest University, Winston-Salem, North Carolina
  - Southern Oregon Orthopedics Research Foundation, Medford, Oregon